CLINICAL TRIAL: NCT05933343
Title: Ethibond Suture Compared to Vessel Loop as Draining Seton for Complex Anal Fistulas; a Multicenter Randomized Clinical Trial
Brief Title: Ethibond Suture vs Vessel Loop as Draining Seton for Complex Anal Fistulas
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit the required number of patients as per the sample size calculated
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Rizkalla, Sameh M.D., Project Scientist, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCF06282023
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ethibond suture (Active Comparator): Patients with complex anal fistula will undergo placement of Ethibond™ 1 suture as a drainage seton
  Interventions: Procedure: Ethibond suture
- Vessel loop (Active Comparator): Patients with complex anal fistula will undergo placement of vessel loop as a drainage seton
  Interventions: Procedure: Vessel loop

INTERVENTIONS:
Procedure: Ethibond suture — An Ethibond™ 1 suture will be placed as a drainage seton for complex anal fistula
  Arms: Ethibond suture
Procedure: Vessel loop — A vessel loop will be placed as a drainage seton for complex anal fistula
  Arms: Vessel loop

SUMMARY:
Drainage seton is usually placed for long-term control of symptoms, and hence it has to be effective in drainage of infection, durable, and comfortable to the patients. The present study assumes that different seton materials would attain different drainage capacities, variable durability and impact on QoL. Therefore, the study aims to compare two commonly used seton materials; Ethibond suture and vessel loop, in the management of CAF in terms of effectiveness in draining infection, percent of seton break and its timing, and change in patients' QoL as measured by a validated questionnaire.

DETAILED DESCRIPTION:
The use of seton as a surgical therapy for fistulous disease has been first described by Hippocrates in 430 BCE. Since then several authors have used either cutting or drainage seton to treat CAF. Different materials have been used as seton, including sutures, stainless steel wires, catheters, cables, silicone, and rubber bands. While the main aim of a drainage seton is to simply drain sepsis and control symptoms in the long term, cutting setons are mainly used for eradiation of the fistula pathology by cutting through the fistula tract and anal sphincter muscles, yet at the cost of an increased risk of fecal incontinence (FI).

As the purpose of a drainage seton is to provide long-term, durable drainage of perineal sepsis and control of symptoms, namely discharge, the seton material can have an impact on its function and durability. A review of the variations in seton types and materials showed that the success rates of suture seton (silk, prolene or nylon suture) are higher than those of Penrose drains and catheters. However, there is a paucity of data on the impact of the seton material on the durability of seton and quality of life (QoL)

Drainage seton is usually placed for long-term control of symptoms, and hence it has to be effective in drainage of infection, durable, and comfortable to the patients. The present study assumes that different seton materials would attain different drainage capacities, variable durability, and impact on QoL. Therefore, the study aims to compare two commonly used seton materials; Ethibond suture and vessel loop, in the management of CAF in terms of effectiveness in draining infection, percent of seton break and its timing, and change in patients' QoL as measured by a validated questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older of either sex who present with CAF will be included. Both cryptoglandular fistulas and fistulas secondary to inflammatory bowel disease (IBD)

Exclusion Criteria:

* Simple anal fistulas
* Fistulas secondary to malignancy or irradiation therapy
* Pregnant women
* Patients with pre-existing setons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Drainage of perianal sepsis | 3 and 12 months
  Change in the perianal disease activity index
Durability | within 12 months
  Incidence and timing of seton break/fall

SECONDARY OUTCOMES:
Quality of life score | 3 and 12 months
  Change in the anal fistula quality of life score which ranges from 14 to 70 and higher values imply greater impact on quality of life
Healing | 12 months
  Complete healing of the anal fistula evidenced by absence of external opening and discharge
Continence state | 12 months
  Change in the Wexner incontinence score which ranges from 0 to 20 and higher values imply more severe fecal incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Wexner, M.D., Study Chair — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No